CLINICAL TRIAL: NCT01575314
Title: Cost-consequence Analysis of Parenchymal Stapling Device Versus Hand-sewing for Pulmonary Lobectomy in Lung Disease: A Randomized Controlled Trial
Brief Title: Cost-consequence Analysis of Parenchymal Stapling Device Versus Hand-sewing for Pulmonary Lobectomy in Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Apichat Tantraworasin, General thoracic surgery unit, Department of Surgery, Faculty of Medicine, Chiang Mai University Hospital, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUR-11-09-26A-13-X
Record Dates: First submitted 2012-04-06; First posted 2012-04-11 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Malignant Neoplasm of Bronchus or Lung, Unspecified
Keywords: stapling device; lobectomy; cost utility
MeSH Terms: interventions — Surgical Staplers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stapling device (Experimental): stapling device refer to patients who were randomized to use stapler for dividing lung parenchyma.
  Interventions: Device: stapling device
- hand sewn (No Intervention): hand sewn refer to patients who were randomized to use hand suturing for dividing lung parenchyma.

INTERVENTIONS:
Device: stapling device — Stapling device include GIA 80, TA 45, endo GIA 60, endo GIA 45
  Other Names: stapler
  Arms: stapling device

SUMMARY:
The purpose of this study is to compare the efficacy and cost difference of using a parenchymal stapling device versus hand sewing for a pulmonary lobectomy in patients with lung disease (mass or others).

DETAILED DESCRIPTION:
There are many lung diseases that need surgical treatment including malignancy lesion or benign lesions such as lung bleb or bullae, lung cyst, benign tumor, infection (necrotizing pneumonia, lung abscess, aspergilloma) etc. One of the most common procedure is pulmonary lobectomy. The surgical method for dividing parenchyma when performing lobectomy was divided in two methods. In the past, the investigators used hand-sewn technique but this procedure was time-consuming, high risk of air leakage, infection and re-operation, long length of hospital stay and high total cost of treatment. In the present time, the investigators use stapling device which has been used worldwide in various field of surgery since 1995. Many studies proved that using stapling devices can reduce post-operative complication, length of hospital stay and total cost of treatment and also became the standard instrument for lung surgery. In Thailand, these devices have been used for at least 5 years but they were not included in all of Health Insurance of Thai Government. Many patients had to pay for these devices by themselves, approximately 323-484.5 USD. Therefore, the investigators try to prove the hypothesis that using stapling devices for lung surgery would reduce the cost of treatment, post-operative air leakage, re-operative rate, length of hospital stay and time of surgery. The result of this study may effect the decision for including these devices in the Health Insurance of Thai Government.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed lung diseases that need to perform pulmonary lobectomy

Exclusion Criteria:

* Patients have complete fissure. therefore, no procedure need to divide the lung parenchyma.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Post-operative air leak, operative time, and duration of air leak | In the operative day, after surgery, until patient can be discharged.
  To compare post-operative air leakage between two groups. This data will be analyzed by fisher exact probability test. We will start observation of the air leakage at postoperative day 1. The stoping role is when statistically significant difference occur. We will measure and report in the number of patients who have post-operative air leakage.

SECONDARY OUTCOMES:
cost of treatment | within the time that patient admit in the hospital
  The cost measurements for each treatment arm focused on the following: 1) direct medical cost (costs of goods and services that are directly provided by the health care system including surgical equipment, drugs and nursing care), 2) direct non-medical cost (costs of goods and services used for health care not directly provided by the heath care system such as transportation, additional meals for patient or their relatives and residence for their relatives),and 3) indirect cost (costs of health care consumption gained as a result of a health care intervention and value of production loss due to illness or treatment such as income lost from sick-leave).
Re-operation due to postoperative air leakage | 8 month after recording data
  To compare the re-operation due to air leakage between two groups. This data will be analyzed by fisher exact probability test. We will record the re-operation due to air leakage. The stopping role is when statistically significant difference occur. In general, we accepted re-operation for air leakage especially patients who have chronic lung disease (COPD), the rate of re-operation that we can accept approximately 20-30 percent We will measure and report in the number of patients who have to perform re-operation due to post-operative air leakage.
Length of Hospital stay | 8 month after recording data
  To compare the length of hospital stay between two groups. Counting of Length of hospital stay (days) will start at 1st post-operative day until discharge. This data will be analyzed by t-test.
  We will measure and report in the unit of time (days).

CONTACTS AND LOCATIONS:
Overall Officials: Apichat Tantraworasin, M.D., Principal Investigator — Department of Surgery, Faculty of medicine, Chiang mai University
Locations (1):
- Department of surgery, Faculty of medicine, Chiang Mai University Hospital, Amphoe Meung, Chaing Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moggi L, Giustozzi GM, Cagini L, Boselli C. [Surgical staplers in thoracic surgery]. G Chir. 1992 Apr;13(4):177-9. Italian. PMID 1637625
- [Derived] Tantraworasin A, Seateang S, Bunchungmongkol N. Staplers versus hand-sewing for pulmonary lobectomy: randomized controlled trial. Asian Cardiovasc Thorac Ann. 2014 Mar;22(3):309-14. doi: 10.1177/0218492313491754. Epub 2013 Aug 19. PMID 24585907
- See also: Click here for more information about this study — http://www.hitap.net